CLINICAL TRIAL: NCT01056367
Title: Resistant Hypertension in Patients With Type-II-Diabetes Mellitus: Prevalence, Characterization and Treatment
Brief Title: Resistant Hypertension in Patients With Type-II-Diabetes Mellitus
Acronym: RESIST
Status: Completed | Type: Observational
Sponsor: Svendborg Hospital (Other)
Responsible Party: Principal Investigator, Trine Koustrup Soender, Medical Doctor, Svendborg Hospital
Other Study IDs: RESIST
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Resistant Hypertension; NIDDM
Keywords: Resistant hypertension; Type-II-Diabetes Mellitus; Arterial stiffness; Ventricular function
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Only serum and plasma samples are used and saved for later analysis.
Oversight: Data Monitoring Committee: No

SUMMARY:
The risk of cardiovascular disease (CVD) in patients with type-II-diabetes mellitus (type-II-DM)is more than doubled and CVD accounts for 70% of deaths in this group of patients.

Hypertension is a major risk factor for CVD in patients with type-II-DM and a major contributor cardiovascular mortality. Uncontrolled- (UH) and resistant hypertension (RH)are more common in patients with type-II-DM, why further bloodpressure (BP) control is needed.

The prevalence of UH and RH has not been examined in a consecutive Danish outpatient population with type-II-DM.

The purpose of this study is to examine the prevalence of resistant hypertension in patients with type-II-diabetes and to examine the characteristics of patients with resistant hypertension as compared to patients with controlled hypertension with regards to arterial stiffness.

DETAILED DESCRIPTION:
The risk of cardiovascular disease (CVD) in patients with type-II- diabetes mellitus (type-II-DM) is more than doubled and CVD accounts for 70% of deaths in this group of patients. Hypertension is a major risk factor for CVD in patients with type-II-DM with a major increase in diabetes-related death as a result. Controlled hypertension as well as uncontrolled- and resistant hypertension is more common in patients with type-II-DM than in the general population and are major contributors to CVD and cardiovascular mortality.

Resistant hypertension is defined as BP above 130 mmHg systolic and / or 80 mmHg diastolic despite treatment with 3 antihypertensive agents or more, of which one should be a diuretic, or controlled BP on four antihypertensive agents or more.

The NHANES study estimated the prevalence of hypertension in patients with type-II-DM to 71% and showed that among those with type-II-DM and hypertension only 31% had controlled BP. It is furthermore estimated that resistant that hypertension is present in up to 30% of a hypertensive population and the ALLHAT trial found that 50% of hypertensives needed treatment with three or more antihypertensive agents.

Type-II-DM promotes both small and large artery disease, whereas hypertension promotes primarily large artery disease. As such type-II-DM and hypertension together may influence the entire vascular system. Type-II-DM is strongly associated with development of heart failure and atherosclerosis and it is therefore important to investigate parameters that reflect arterial stiffness (AS), left ventricular function and degree of atherosclerosis.

AS is an age dependent process, where the arterial wall degenerate and elastic fibers are replaced by collagen fibers. The process is accelerated by cardiac risk factors and increased AS can be regarded as both an individual risk factor and a marker reflecting atherosclerosis.

AS can be estimated by pulse wave analysis (PWA) including pulse wave velocity (PWV).

As blood is pumped out of the heart, a pulse wave is created. The pulse wave propagates along the vessels and is reflected from the arterial wall at sites of increased impedance. In healthy elastic arteries the reflected wave reaches the aorta during diastole resulting in increased coronary perfusion. In stiff arteries the reflected wave propagates faster and reaches the aorta during systole before closure of the aortic valve, thereby increasing pulse pressure, systolic pressure and reducing diastolic pressure and thereby coronary perfusion.

Augmentation Index (AIx) measured using PWA is related to ischemic heart disease (IHD) risk factors, among other hypertension and diabetes, and is an independent predictor of mortality in patients with IHD. It is therefore important to examine the relationship between BP and AS, as it may characterize the patients with uncontrolled and resistant hypertension.

A consequence of increased AS is left ventricular hypertrophy (LVH) and a common echocardiographic finding in patients with hypertension, type-II-DM and LVH, is diastolic dysfunction. This is often seen before the onset of systolic dysfunction and any symptoms of CVD.

Coronary artery calcium (CAC) score is closely related to atherosclerosis and is a number reflecting the degree and extent of calcium deposits in the walls of the coronary arteries, as demonstrated by cardiac computed tomography. CAC score represents overall plaque burden and is also an independent predictor of cardiovascular events (CVE) and cardiovascular death in asymptomatic patients. In patients with type-II-DM the extent of CAC score is similar to that of patients with coronary artery disease (CAD). Measurement of CAC score can be used as advanced risk assessment. As CAC score is high in patients with cardiac risk factors it is possible that CAC score is reduced when minimizing cardiac risk factors.

The relationship between BP, AS and left ventricular function score may provide further methods of risk stratification and new strategies for treatment of uncontrolled and resistant hypertension in patients with type-II-DM.

Hypothesis

1. Uncontrolled and resistant hypertension is present in more than 50% of consecutive patients with type-II-DM in an out-patient clinic.
2. Increased AS, diastolic dysfunction and high CAC score are more common in patients with type-II-DM with uncontrolled or resistant hypertension than in patients with controlled BP.
3. AS, diastolic function and CAC are improved with increased control of BP.

To test these hypotheses we wish to conduct two studies:

1. A descriptive study in which the prevalence of uncontrolled and resistant hypertension in consecutive out-patients with type-II-DM is assessed.
2. Assessment of AS, diastolic function and CAC in patients with type-II-DM with uncontrolled and resistant hypertension and the changes in these parameters during intensified treatment. This is compared to patients with controlled BP.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years, informed consent, hypertension, type-II-diabetes mellitus

Exclusion Criteria:

* Non-compliance, s-creatinin above 200, AFli

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from diabetic outpatient clinic
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pulse wave velocity | one year

SECONDARY OUTCOMES:
Myocardial contractility | One year
Pulse wave analysis | One year

CONTACTS AND LOCATIONS:
Overall Officials: Trine K Sønder, Cand.med., Principal Investigator — Department of Medical Research, Svendborg Hospital
Locations (1):
- Department of Medical Research, Svendborg Hospital, Svendborg, Denmark